CLINICAL TRIAL: NCT05918536
Title: Orthopedic Oncology Surgery: Navigation, Intraoperative Imaging and Virtual Reality
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Regina Elena Cancer Institute (Other)
Collaborators: Azienda Policlinico Umberto I (Other); I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: RS1686/22
Record Dates: First submitted 2023-03-28; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Neoplasms; Muscle Neoplasm
MeSH Terms: conditions — Neoplasms; Muscle Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Popolation
  Interventions: Diagnostic Test: evaluate the quality of surgical margins achievable with the use of navigated Intraoperative CT

INTERVENTIONS:
Diagnostic Test: evaluate the quality of surgical margins achievable with the use of navigated Intraoperative CT — Noninterventional, prospective study of patients operated on for musculoskeletal neoplasms designed to evaluate the quality of surgical margins achievable with the use of navigated Intraoperative CT

SUMMARY:
Noninterventional, prospective study of patients operated on for musculoskeletal neoplasms designed to evaluate the quality of surgical margins achievable with the use of navigated Intraoperative CT

ELIGIBILITY:
Inclusion Criteria:

* Age: no limit
* Patients with musculoskeletal neoplasms predominantly in complex sites
* Patients who will have to undergo surgical resection/amputation for the management of their clinical case
* Preparation of preoperative planning discussed at DMT
* Surgery performed with the aid of Intraoperative CT Navigated
* Written informed consent

Exclusion Criteria:

- Inability to perform pre-post treatment assessment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with primary and secondary cancers of the musculoskeletal system with estimated survival greater than one year who are candidates for bone resection surgery or wide excision of soft tissue lesion and/or radio and chemotherapy treatments
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2022-05-17 (Actual); Primary Completion 2025-05-17 (Estimated); Study Completion 2025-11-17 (Estimated)

PRIMARY OUTCOMES:
Quality of life | Baseline
  To evaluate the quality of the Surgical Margin in terms of the percentage of oncologically adequate resections, in patients with Musculoskeletal neoplasms undergoing navigated resection surgery with Intraoperative CT

CONTACTS AND LOCATIONS:
Locations (1):
- "Regina Elena" National Cancer Institute, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided